CLINICAL TRIAL: NCT02813057
Title: Quantitative Assessment of the Impacts of Stoppa Repair and Total Extraperitoneal Repair on the Lower Extremity Muscular Functions in Cases of Unilateral Inguinal Hernia; a Randomized Controlled Study
Brief Title: Impacts of Stoppa and Total Extraperitoneal Inguinal Hernia Repair on the Lower Extremity Muscular Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201203
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stoppa repair (Active Comparator): Stoppa inguinal hernia repair
  Interventions: Procedure: Stoppa inguinal hernia repair
- TEP repair (Experimental): Total extraperitoneal inguinal hernia repair
  Interventions: Procedure: Total extraperitoneal inguinal hernia repair

INTERVENTIONS:
Procedure: Stoppa inguinal hernia repair — Stoppa inguinal hernia repair
  Arms: Stoppa repair
Procedure: Total extraperitoneal inguinal hernia repair — Total extraperitoneal inguinal hernia repair
  Arms: TEP repair

SUMMARY:
Comparison of physical activity parameters of the lower extremity muscles in patients who received total extraperitoneal repair (TEP) and STOPPA repair.

DETAILED DESCRIPTION:
The patients were evaluated during the preoperative period and in the postoperative day 3, to achieve an isometric and isokinetic, objective assessment of the pain-related lower extremity muscular function changes.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral inguinal hernia

Exclusion Criteria:

* Contralateral hernia repair history
* Recurrent inguinal hernia
* Incarceration or strangulation
* Bilateral inguinal hernia
* Severe congestive heart failure
* Severe hypertension
* Rheumatoid arthritis
* Systemic or neurologic diseases altering lower extremity functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Functional loss in lower extremity muscles | postoperative day 3
  Physical activity parameters (isokinetic and isometric values) of the lower extremity muscular functions were measured with a dynamometer.

SECONDARY OUTCOMES:
Duration of hospital stay | From time of admission to time of discharge an approximate length of three days
Postoperative pain score | Postoperative 12 hour
  Visual analog score assessment of post operative pain
Recurrence rate | Postoperative 4 months
  Number of patients with recurrence
Complications | Postoperative 1 month
  Complications like infection, seroma, hematoma, abscess, wound healing problems and urinary retension.

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan Mesci, Assoc. Prof., Study Director — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akgul N, Yaprak M, Dogru V, Balci N, Arici C, Mesci A. Quantitative assessment of the impacts of stoppa repair and total extraperitoneal repair on the lower extremity muscular functions in cases of unilateral inguinal hernia: a randomized controlled study. Hernia. 2017 Jun;21(3):377-382. doi: 10.1007/s10029-016-1559-6. Epub 2016 Dec 10. PMID 27942876